CLINICAL TRIAL: NCT03238131
Title: Comparison of Ivermectin Alone With Albendazole (ALB) Plus Ivermectin (IVM) in Their Efficacy Against Onchocerciasis
Brief Title: IVM Alone vs ALB + IVM Against Onchocerciasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Professor of International Health, Medicine and Pathology, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-11-36
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Onchocerciasis
MeSH Terms: conditions — Onchocerciasis | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IVM annually (standard treatment) (Active Comparator): The comparator (standard treatment) IVM 200 µg/kg body weight given at 0, 12 and 24 months plus vitamin pills at 6 and 18 months.
  Interventions: Drug: Ivermectin
- IVM plus ALB twice annually (Experimental): IVM 200 µg/kg plus ALB 800 mg (regardless of weight) given at 0, 6, 12, 18, 24 months
  Interventions: Drug: Ivermectin; Drug: Albendazole
- IVM plus ALB once annually (Active Comparator): IVM 200 µg/kg plus ALB 800 mg given at 0, 12, 24 months plus vitamin pills at 6 and 18 months.
  Interventions: Drug: Ivermectin; Drug: Albendazole
- IVM twice annually (Active Comparator): IVM 200 µg/kg given 0, 6, 12, 18, and 24 months
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Participants are either given Ivermectin alone or Ivermectin in combination with Albendazole
Drug: Albendazole — Albendazole will be given to participants in Arm 2 and 3 in combination with Ivermectin at varying time points.
  Arms: IVM plus ALB once annually; IVM plus ALB twice annually

SUMMARY:
Onchocerciasis is a vector-borne nematode parasitic disease that causes severe disability. Onchocerciasis affects approximately 33 million people, mostly in 30 countries in sub-Saharan Africa (with small foci in Latin America and Yemen) 1This disease causes blindness and severe skin disease and it is spread by black flies. O. volvulus adult worms live in subcutaneous nodules. O. volvulus adult worms are larger and less sensitive to available drug treatments than those of the species that cause Lymphatic Filariasis (LF). They also have a longer lifespan (approximately 14 years rather than the estimated 7 years for LF parasites). Several programs and developments have greatly improved the Onchocerciasis. situation since the 1970's when the Onchocerciasis Control Programme (OCP) in West Africa (green countries in the map) was initiated. OCP relied exclusively on vector (black fly) control in its early years. However, following the appearance of Ivermectin (Mectizan) on the scene in the late 1980's, OCP transitioned to become a drug distribution program with annual IVM MDA in 11 countries. OCP ended in 2002. This was replaced by the African Program for Onchocerciasis Control (APOC) which coordinates community directed distribution of IVM MDA in 28 African countries (including the former OCP countries). OCP and APOC have done a good job of reducing parasite infection intensities and Onchocerciasis disease rates in many endemic countries. Unfortunately, there is no real end in sight for the APOC approach (apart from a funding endpoint in 2015); while it may be possible to eliminate Onchocerciasis. In selected areas by MDA with IVM (alone, or combined with vector control), disease control programs in most African countries will require active maintenance for many years to come. While IVR has good activity against the parasite larvae that cause disease in the skin and eye (microfilariae or Mf), it does not kill O. volvulus adult worms, and they resume production of Mf that can lead to transmission of new Onchocerciasis. Cases by black flies after a few months. APOC activities are focused on areas with high infection rates (where disease risks are highest). However, extensive areas in Africa where fewer than 20% of adult men have Onchocerciasis nodules detectable by palpation are not receiving interventions for Onchocerciasis at this time. These areas are not disease free. (Onchocerciasis dermatitis can be severe in hypoendemic areas), and they also may serve as a source for reintroduction of the parasite into previously controlled areas after interventions stop.

DETAILED DESCRIPTION:
Onchocerciasis control programs have relied on annual MDA with IVM at a dose of 150-200 µg/kg. This regimen kills skin (and eye) Mf, thereby reducing disease and (in some areas) transmission. However, standard IVM monotherapy has little macrofilaricidal activity against adult O. volvulus, and it does not permanently sterilize adult worms, which have a reproductive life span of 12-14 years. More effective drugs or dosing schedules that have embryo-static or macrofilaricidal activity could drastically reduce the number of years required to interrupt transmission of Onchocerciasis. IVM has activity against adult O. volvulus when it is given at high doses four times per year for several years. This regimen caused some adverse events, and is not practical for national control programs. By contrast, whereas ALB has little effect on O. volvulus Mf, the drug has embryo-toxic effects at standard doses manifest as partial suppression (by 66%) of skin Mf counts for at least one year. ALB given at doses of 800 mg produced a more sustained reduction in Mf relative to a dose of 400 mg, but higher doses did not improve efficacy. It is not known whether ALB produces transient or permanent female worm sterility. Administration of a single 400 mg dose of ALB combined with IVM 200 µg/kg failed to a show greater reduction in Mf or macrofilaricidal activity compared to IVM alone; however, combination therapy suppressed embryogenesis more than IVM alone. These studies involved small numbers of participants, used ALB only at a dose of 400 mg, and followed the participants for just one year. Thus, IVM combined with ALB at higher doses given more than once per year may generate more sustained reduction in Mf by reducing female fertility or by killing adult worms.

IVM and ALB are very safe and highly effective anti-filarial drugs when given singly or in combination.

ALB causes degenerative alterations in the tegument and intestinal cells of the worm by binding to the colchicine-sensitive site of tubulin, thus inhibiting its polymerization or assembly into microtubules. The loss of cytoplasmic microtubules leads to impaired uptake of glucose by larval and adult stages of the parasite, and depletes glycogen stores. Degenerative changes in endoplasmic reticulum and mitochondria of the germinal layer, and the subsequent release of lysosomal enzymes result in decreased production of adenosine triphosphate, which is the source of energy required for survival of the helminth. Due to diminished energy production, the parasite is immobilized and eventually dies. The drug has been shown to cause occasionally (<1% of treated patients) reversible reductions in total white blood cell count. It has also been associated with slight increases in liver transaminases in ~16% of patients. The enzymes return to normal levels with cessation of treatment. These abnormalities are associated primarily with prolonged treatment for such diseases as neurocysticercosis and hydatid diseases, not single dose treatment which is being proposed here. ALB given with fatty foods as proposed in the current protocol will increase absorption and may increase the risk of adverse side effects.

IVMis an avermectin compound of macrocyclic lactones derived from the bacterium Streptomyces avermitilis. The mechanism by which IVM kills LF microfilariae is not known with certainty, but the drug interferes with glutamate gated ion channels that can affect parasite contractility and release of immunomodulatory molecules by the parasite. IVM also has a direct effect on the central nervous system and muscle function as it enhances strength of inhibitory neurotransmission pathways. The main concern with use of IVM in animals and humans is neurotoxicity, which can be manifest as ataxia. Neurotoxicity has not been observed in humans given single dose IVM for LF or other parasitic infections, and the drug has been used to treat millions of people with LF and Onchocerciasis. Peak IVM serum concentrations are reached approximately 4-5 hours after administration. The half-life of IVM in various populations ranges from 12 to 56 hours 12. There is no evidence of drug:drug interaction between ALB and IVM.

IVM can cause nausea, dizziness and occasionally pruritus, but these are infrequent, transient and usually mild. Major side effects occur with heavy infections of Loa loa; however, this parasite is not endemic in Ghana.

In Ghana the chiefs and elders are the custodians of the land so they must first to be contacted for permission to enter their communities. The study objectives and procedures are then explained to them, and if they accept it then the research team is allowed to enter the communities to explain the research aims and procedures to their subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-60 years residing in Ashanti and Central Region of Ghana
* ≥1 accessible nodules
* any Mf/mg based on skin snips
* Willingness to give informed consent to participation in the study

Exclusion Criteria:

* Last IVM treatment < 7 months
* Pregnant (do pregnancy test) + breastfeeding
* Permanent disability, serious medical illnesses such as a stroke, advanced heart disease, uncontrolled diabetes, emphysema, etc that prevents or impedes study participation and/or comprehension
* Weight of <40kg suggesting malnourishment
* AST/ALT, γ-GT > 1.5 upper limit of normal
* Significant glycosuria or proteinuria (2+ or 3+ protein or glucose)
* Any one or more of the previous criteria is sufficient to exclude study participation
* Not willing or able to give informed consent to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The percent fertile female O.volvulus worms in nodules | 36 months
  Total number of live versus dead female worms in nodules

SECONDARY OUTCOMES:
Percent reduction in skin Mf/mg | 0 months
  Percent of live female worms in nodules
Percent reduction in skin Mf/mg | 6 months
  Total number of live versus dead female worms in nodules compared to time point zero
Percent reduction in skin Mf/mg | 18 months
  Total number of live versus dead female worms in nodules compared to time point zero
Percent reduction in skin Mf/mg | 36 months
  Total number of live versus dead female worms in nodules compared to time point zero
Number of nodules with intact Mf | 36 months
  number of nodules with intact Mf at 36 months following initial therapy
Soil Transmitted Helminth (STH) infections | 36 months
  Assessment of the different treatment regimens on STH infections based on presence of intensity of ova in stools.

CONTACTS AND LOCATIONS:
Locations (1):
- Committee on Human Research Publications and Ethics, Kumasi, Ashanti Region, Ghana

REFERENCES:
- [Background] Basanez MG, Pion SD, Churcher TS, Breitling LP, Little MP, Boussinesq M. River blindness: a success story under threat? PLoS Med. 2006 Sep;3(9):e371. doi: 10.1371/journal.pmed.0030371. PMID 17002504
- [Background] Gardon J, Boussinesq M, Kamgno J, Gardon-Wendel N, Demanga-Ngangue, Duke BO. Effects of standard and high doses of ivermectin on adult worms of Onchocerca volvulus: a randomised controlled trial. Lancet. 2002 Jul 20;360(9328):203-10. doi: 10.1016/S0140-6736(02)09456-4. PMID 12133654
- [Background] Zahner H, Schares G. Experimental chemotherapy of filariasis: comparative evaluation of the efficacy of filaricidal compounds in Mastomys coucha infected with Litomosoides carinii, Acanthocheilonema viteae, Brugia malayi and B. pahangi. Acta Trop. 1993 Jan;52(4):221-66. doi: 10.1016/0001-706x(93)90010-9. PMID 8094587
- [Background] Awadzi K, Hero M, Opoku O, Buttner DW, Gilles HM. The chemotherapy of onchocerciasis. XV. Studies with albendazole. Trop Med Parasitol. 1991 Dec;42(4):356-60. PMID 1796233
- [Background] Awadzi K, Addy ET, Opoku NO, Plenge-Bonig A, Buttner DW. The chemotherapy of onchocerciasis XX: ivermectin in combination with albendazole. Trop Med Parasitol. 1995 Dec;46(4):213-20. PMID 8826100
- [Background] Awadzi K, Edwards G, Duke BO, Opoku NO, Attah SK, Addy ET, Ardrey AE, Quartey BT. The co-administration of ivermectin and albendazole--safety, pharmacokinetics and efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2003 Mar;97(2):165-78. doi: 10.1179/000349803235001697. PMID 12803872
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686
- [Background] Horton J. Albendazole: a broad spectrum anthelminthic for treatment of individuals and populations. Curr Opin Infect Dis. 2002 Dec;15(6):599-608. doi: 10.1097/00001432-200212000-00008. PMID 12821837
- [Background] Geary TG. Ivermectin 20 years on: maturation of a wonder drug. Trends Parasitol. 2005 Nov;21(11):530-2. doi: 10.1016/j.pt.2005.08.014. Epub 2005 Aug 26. PMID 16126457
- [Background] Moreno Y, Nabhan JF, Solomon J, Mackenzie CD, Geary TG. Ivermectin disrupts the function of the excretory-secretory apparatus in microfilariae of Brugia malayi. Proc Natl Acad Sci U S A. 2010 Nov 16;107(46):20120-5. doi: 10.1073/pnas.1011983107. Epub 2010 Nov 1. PMID 21041637
- [Background] Awadzi K, Edwards G, Opoku NO, Ardrey AE, Favager S, Addy ET, Attah SK, Yamuah LK, Quartey BT. The safety, tolerability and pharmacokinetics of levamisole alone, levamisole plus ivermectin, and levamisole plus albendazole, and their efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2004 Sep;98(6):595-614. doi: 10.1179/000349804225021370. PMID 15324466
- [Background] Kitzman D, Wei SY, Fleckenstein L. Liquid chromatographic assay of ivermectin in human plasma for application to clinical pharmacokinetic studies. J Pharm Biomed Anal. 2006 Mar 3;40(4):1013-20. doi: 10.1016/j.jpba.2005.08.026. Epub 2005 Oct 19. PMID 16242280
- [Background] Cringoli G, Rinaldi L, Maurelli MP, Utzinger J. FLOTAC: new multivalent techniques for qualitative and quantitative copromicroscopic diagnosis of parasites in animals and humans. Nat Protoc. 2010 Mar;5(3):503-15. doi: 10.1038/nprot.2009.235. Epub 2010 Feb 25. PMID 20203667